CLINICAL TRIAL: NCT00833560
Title: Clinical Study on Induction of Remission Using Bortezomib (Vel), Cyclophosphamide (C), and Dexamethasone (D) in Patients Until 60 Years of Age With Untreated Multiple Myeloma and Planned for a High Dose Chemotherapy: (VelCD; Deutsche Studiengruppe Multiples Myelom [DSMM] XIa)
Brief Title: A Study of Bortezomib, Cyclophosphamide, and Dexamethasone in Patients With Untreated Multiple Myeloma and Planned for a High Dose Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005242; 26866138MMY2031 (Other: Janssen-Cilag G.m.b.H, Germany); 2005-003902-27 (EudraCT Number)
Record Dates: First submitted 2009-01-23; First posted 2009-02-02 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Untreated multiple myeloma; Bortezomib; VELCADE; Cyclophosphamide; Dexamethasone; Chemotherapy; Remission therapy; Induction therapy; Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclophosphamide + Bortezomib + Dexamethasone (Experimental): Part 1 will be the dose titration part for cyclophosphamide. Participants will receive cyclophosphamide, bortezomib, and dexamethasone for 3 cycles. In Part 2, participants will receive cyclophosphamide (dose determined in Part 1) with pre-defined dose of bortezomib and dexamethasone for 3 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — In Part 1, cyclophosphamide with dose ranging from 900 to 1500 mg will be administered intravenously on Day 1 of each 21 day cycle for 3 cycles to determine optimal dose. In Part 2, optimal dose determined in Part 1 will be administered on Day 1 of each 21 day cycle for 3 cycles.
Drug: Bortezomib — Bortezomib 1.3 mg/m2 will be administered intravenously on Days 1,4,8, and 11 of each 21 day cycle for 3 cycles in both parts (Part 1 and Part 2).
  Other Names: VELCADE
Drug: Dexamethasone — Participants will receive dexamethasone 40 mg orally or intravenously on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21 day cycle for 3 cycles in both parts (Part 1 and Part 2).

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of bortezomib in combination with a standard regimen of cyclophosphamide and dexamethasone.

DETAILED DESCRIPTION:
This is open-label (both the participant and the investigator know what treatment participants will receive), prospective (participants are identified and then followed forward in time for the outcome of the study), multi-centre, and non-randomized (participants are assigned to different treatment groups by the investigator) study. The study will be conducted into 2 parts (Part 1 and Part 2). Approximately 400 participants will be enrolled (30 in Part 1 and 370 in Part 2). In Part 1 the optimum dose of cyclophosphamide will be evaluated and in Part 2 the selected dose of cyclophosphamide from Part 1 will be administered. Part 2 will include a screening period of a maximum of 14 days followed by chemotherapy (bortezomib, cyclophosphamide, and dexamethasone) of a maximum of three 21-day cycles. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, electrocardiogram, and clinical laboratory tests which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically diagnosed with multiple myeloma stage II/III
* Participants without preceding cytostatic (tending to retard cellular activity and multiplication) treatment (pretreatment with radiation or dexamethasone is allowed)
* Agree to use one of the contraception methods as defined in the protocol
* Karnofsky performance status 60 percent or more
* Adequate laboratory test values

Exclusion Criteria:

* Non-secretory multiple myeloma
* Estimated life expectancy less than 3 months
* History of cancer (except basal cell carcinoma) in the last 5 years
* Peripheral neuropathy (disorder of the peripheral nerves) grade 2 or more
* Positive human immunodeficiency virus test and active hepatitis B and/or hepatitis C
* Pregnant or breast-feeding female participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (34):
- Germany (34):
  - Berg
  - Berlin
  - Bremen
  - Dresden
  - Erlangen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Halle
  - Hamburg
  - Hamm
  - Hanover
  - Homburg
  - Jena
  - Karlsruhe
  - Kiel
  - Lübeck
  - Magdeburg
  - Mainz
  - Mutlangen
  - München
  - Münster
  - Nuremberg
  - Oldenburg
  - Potsdam
  - Regensburg
  - Rehling
  - Rostock
  - Stuttgart
  - Tübingen
  - Ulm
  - Villingen-Schwenningen
  - Würzburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 401 participants were enrolled at 41 study sites in Germany.
Pre-assignment Details: Out of 401 participants, 399 participants were treated in both the Parts. Out of 399 participants, 395 participants were evaluated as 4 participants who had received cyclophophamide dose of greater than 1350 mg/m^2 per cycle in Part 1 were excluded.
Groups:
- Cyclophosphamide + Bortezomib + Dexamethasone: Cyclophosphamide + Bortezomib + Dexamethasone for three 21-day cycles
Period: Overall Study
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Started | 395
Completed | 353
Not Completed | 42
Not completed — Toxicity | 13
Not completed — Adverse Event | 11
Not completed — Protocol Violation | 6
Not completed — Lack of Efficacy | 4
Not completed — Death | 2
Not completed — Pregression of other disease | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Number analyzed (Participants) | 395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (6.5)
Age, Customized [Number; unit: Participants]
  Between 20 and 39 years | 17
  Between 40 and 49 years | 109
  Between 50 and 60 years | 253
  >65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 229

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complete Response (CR) + Partial Response (PR) (Efficacy Set)
Description: CR and PR are defined by the local investigator according to the current European Group for Blood and Marrow Transplantation (EBMT) criteria. According to EBMT criteria, CR is defined as the absence of serum and urine monoclonal paraprotein + no increase in size or number of lytic bone lesions; and PR is defined as not all CR criteria + 50 percentage or more reduction in serum monoclonal paraprotein.
Time Frame: Up to Day 63
Population: Efficacy analysis set: Participants of the safety analysis set (who received bortezomib at least once independently of accordance to the protocol) who had an evaluable investigator based assessment of success of therapy at the end of study visit (ie, assessment by local investigator as CR, PR, minimal response, stable disease, progressive disease).
Measure: Number; unit: Participants
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Number analyzed (Participants) | 391
Participants | 334
Statistical Analysis 1: Comparison: Cyclophosphamide + Bortezomib + Dexamethasone; Test type: Superiority or Other; p < 0.0001, Two - sided binomial test; Percentage of participants with response = 85.4, 95% CI 2-sided [81.5 to 88.8]

2. Secondary Outcome: Participants With Complete Response (CR) + Partial Response (PR) (Per-protocol Analysis Set)
Description: as for outcome 1
Time Frame: Up to Day 63
Population: Per-protocol analysis set: It includes the participants who completed the entire clinical study without major protocol violations.
Measure: Number; unit: Participants
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Number analyzed (Participants) | 324
Participants | 284
Statistical Analysis 1: Comparison: Cyclophosphamide + Bortezomib + Dexamethasone; Test type: Superiority or Other; p < 0.0001, Two-sided binomial test; Percentage of participants with response = 87.7, 95% CI 2-sided [83.6 to 91.0]

3. Secondary Outcome: Percentage of Participants With Complete Response + Partial Response in Relation to Cytogenetic Subgroups (Efficacy Set)
Description: Response rate was defined as the percentage of participants with response of combined CR+PR according to the EBMT criteria. As per the EBMT criteria, CR is defined as the absence of serum and urine monoclonal paraprotein and no increase in size or number of lytic bone lesions; PR is defined as not all CR criteria and 50 percentage or more reduction in serum monoclonal paraprotein. Percentage of participants with complete or partial response that carried the indicated cytogenetic marker is reported. Same participant could count in more than one category due to multiple responses possible
Time Frame: Up to Day 63
Population: Efficacy analysis set. N (number of participants analyzed) signifies participants with complete or partial response. "n" signifies number of participants who were evaluable for each specified category (participants that carried the indicated cytogenetic marker).
Measure: Number; unit: Percentage of participants
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Number analyzed (Participants) | 334
Percentage of participants
  13q- (n=112) | 90.2
  t (4;14) (n=38) | 89.5
  17p- (n=31) | 74.2
  Other (n=104) | 87.5
  No changes (n=102) | 84.3

4. Secondary Outcome: Percentage of Participants With Complete Response + Partial Response in Relation to Cytogenetic Subgroups (Per-protocol Set)
Description: as for outcome 3
Time Frame: Up to Day 63
Population: Per-protocol analysis set. N (number of participants analyzed) signifies participants with complete or partial response. "n" signifies number of participants who were evaluable for each specified category (participants that carried the indicated cytogenetic marker).
Measure: Number; unit: Percentage of participants
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Number analyzed (Participants) | 284
Percentage of participants
  13q- (n=92) | 92.4
  t (4;14) (n=34) | 91.2
  17p- (n=24) | 87.5
  Other (n=87) | 88.5
  No changes (n=87) | 85.1

ADVERSE EVENTS:
Time Frame: From date of inform consent signed to 30 days after the last bortezomib dosing or, if earlier, until start of an alternative myeloma therapy.
Arm/Group | Cyclophosphamide + Bortezomib + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 103/395
Other Adverse Events (participants affected / at risk) | 392/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide + Bortezomib + Dexamethasone (N=395)
Pneumonia (Infections and infestations) | 15 (16)
Herpes zoster (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Bacterial sepsis (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Encephalitis herpes (Infections and infestations) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 14 (15)
Disease progression (General disorders) | 3 (3)
Asthenia (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 11 (12)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 2 (2)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 4 (4)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood immunoglobulin G increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Presbyacusis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide + Bortezomib + Dexamethasone (N=395)
Oedema peripheral (General disorders) | 79 (105)
Fatigue (General disorders) | 76 (85)
Pyrexia (General disorders) | 56 (70)
Asthenia (General disorders) | 41 (46)
Oedema (General disorders) | 28 (32)
Pain (General disorders) | 28 (33)
Paraesthesia (Nervous system disorders) | 63 (75)
Headache (Nervous system disorders) | 54 (62)
Polyneuropathy (Nervous system disorders) | 51 (68)
Dizziness (Nervous system disorders) | 48 (55)
Hypoaesthesia (Nervous system disorders) | 27 (30)
Dysgeusia (Nervous system disorders) | 20 (20)
Nasopharyngitis (Infections and infestations) | 47 (50)
Rhinitis (Infections and infestations) | 30 (31)
C-reactive protein increased (Investigations) | 39 (47)
Weight increased (Investigations) | 38 (43)
Haemoglobin decreased (Investigations) | 28 (73)
Alanine aminotransferase increased (Investigations) | 22 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (56)
Bone pain (Musculoskeletal and connective tissue disorders) | 32 (34)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (38)
Night sweats (Skin and subcutaneous tissue disorders) | 36 (39)
Erythema (Skin and subcutaneous tissue disorders) | 28 (31)
Rash (Skin and subcutaneous tissue disorders) | 22 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (49)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (31)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (21)
Sleep disorder (Psychiatric disorders) | 46 (53)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (30)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (27)
Hypertension (Vascular disorders) | 28 (33)
Leukopenia (Blood and lymphatic system disorders) | 211 (680)
Thrombocytopenia (Blood and lymphatic system disorders) | 129 (277)
Anaemia (Blood and lymphatic system disorders) | 77 (132)
Neutropenia (Blood and lymphatic system disorders) | 32 (53)
Nausea (Gastrointestinal disorders) | 105 (141)
Constipation (Gastrointestinal disorders) | 86 (98)
Diarrhoea (Gastrointestinal disorders) | 73 (88)
Vomiting (Gastrointestinal disorders) | 50 (63)
Flatulence (Gastrointestinal disorders) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days